CLINICAL TRIAL: NCT02244996
Title: Cone Rescue in Retinitis Pigmentosa by the Treatment of Lycium Barbarum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Henry HL Chan, PhD, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01121876
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-01

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis pigmentosa; Lycium barbarum; Antioxidation; Visual field; Electroretinogram
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — lycium barbarum polysaccharide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lycium Barbarum (Experimental): Daily Lycium Barbarum dosage: 10g of granules for 12 months
  Interventions: Dietary Supplement: Lycium Barbarum
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lycium Barbarum — Traditional Chinese Herbs
  Other Names: Wolfberry
  Arms: Lycium Barbarum
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Objectives: To study the immediate effect and the persistent effect of Lycium barbarum (LB) treatment on retinal functions, especially the cone function, and retinal structure in patients with retinitis pigmentosa (RP) Design: Randomised controlled double-masked trial

Setting: Primary Care clinical trial

Participants: 120 RP subjects will be recruited from Ophthalmology department at The University of Hong Kong and the Retina Hong Kong. Interventions: Subjects will be randomly allocated to LB (treated with LB granules) or control (treated with placebo) groups for 1 year. After the 1st year, both groups will stop the treatment and all subjects will also have the same eye exam in 6-month period for the 2nd year.

Main outcome measures: The primary outcome is the total sensitivity scores of 30-2 & 60-4 programmes of Humphrey Visual Field Analysis (HVFA). The secondary outcomes are the b-wave amplitudes of Full-field Electroretinogram (ffERG) responses, the amplitudes of direct component and induced component of Multifocal Electroretinogram (mfERG), and the ETDRS visual acuity.

DETAILED DESCRIPTION:
The study was a randomized controlled trial with a double-masked, placebo-controlled design. All the subjects were randomly allocated into either LB (treatment) group or placebo (control) group.

All the eligible subjects had the eye examination, including VA using the Early Treatment of Diabetic Retinopathy Study (ETDRS) chart, refractions, tonometry, external and internal ocular health assessments, and fundus photo-documentation. Three additional tests were conducted to investigate the functional and structural changes in the RP patients, including Ganzfeld Electroretinogram, Humphrey Visual Field Analyser (Zeiss, Dublin, USA) and Spectral-domain Optical Coherent Tomography (SD-OCT) (Heidelberg Engineering, USA).

ELIGIBILITY:
Inclusion Criteria:

Ocular conditions:

* Retinitis pigmentosa;
* best corrected VA LogMAR 0.20 or better;
* Humphrey Visual Field Analysis (HVFA) 30-2 total mean defect > or = 250 Decibel;
* Intra-ocular pressure (IOP) <21 mmHg;
* van Herrick ratio < or = 0.5;
* no other ocular diseases

Dietary conditions:

* Fruit and vegetable intake <10 servings/day;
* spinach or kale intake < or = serving/day;
* dietary lutein intake < or = 5.4mg/day;
* no intake of cod liver oil or omega-3 capsules;
* dietary Lycium barbarum intake < or =10 fruits/week;
* supplement intake < or = 5000 IU/day of Vit. A and < or = 30 IU/day of Vit. E;
* alcoholic consumption < or = 3 beverages/day

Exclusion Criteria:

* BMI > 40;
* intake of any anticoagulants (especially Warfarin),
* pregnant or planning to be pregnant;
* smoking;
* other clinically significant systemic diseases, eg. diabetes, liver disease and heart disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry HL Chan, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Chan HH, Lam HI, Choi KY, Li SZ, Lakshmanan Y, Yu WY, Chang RC, Lai JS, So KF. Delay of cone degeneration in retinitis pigmentosa using a 12-month treatment with Lycium barbarum supplement. J Ethnopharmacol. 2019 May 23;236:336-344. doi: 10.1016/j.jep.2019.03.023. Epub 2019 Mar 12. PMID 30877066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from a retinal disease patient association, Retina Hong Kong, and the Optometry Clinic at The Hong Kong Polytechnic University
Pre-assignment Details: All the eligible subjects had the eye examination, including VA (ETDRS) charts, refractions, tonometry, external and internal ocular health assessments, fundus photo-documentation, Ganzfeld Electroretinogram, Humphrey Visual Field Analyser and Spectral-domain Optical Coherent Tomography
Period: Overall Study
Arm/Group | Lycium Barbarum | Placebo
Started | 25 | 25
Completed | 23 | 19
Not Completed | 2 | 6
Not completed — Lack of Efficacy | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lycium Barbarum | Placebo | Total
Number analyzed (Participants) | 23 | 19 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (12.2) | 48.4 (9.3) | 49.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 9 | 5 | 14
Region of Enrollment [Number; unit: participants]
  Hong Kong | 23 | 19 | 42

OUTCOME MEASURES:

1. Primary Outcome: ETDRS Visual Acuity (High Contrast)
Description: The high contrast visual acuity will be measured at the time point of baseline and 12 months. Visual acuity is to measure the eye's ability to resolve fine detail with full refractive error correction.
  The change of acuity (sec of arc) between 12-month time point and baseline will be provided to show the effect of interventions.
  The changes of the treatment group will be compared with the changes of the placebo group to illustrate the treatment effect of Lycium Barbarum.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: log unit
Arm/Group | Lycium Barbarum | Placebo
Number analyzed (Participants) | 23 | 19
log unit | -0.02 (0.09) | 0.11 (0.17)

2. Secondary Outcome: Visual Field Sensitivity
Description: Humphrey Visual Field Analyser will be used to measure the brightness sensitivity across the central 30 degree visual field at time point of baseline and 12 months. Visual field is to measure the size of the field of view and the sensitivity of the corresponding locations of the field of view.
  The change of sensitivity (dB) between 12-month time point and baseline will be provide to show the effects of interventions.
  The changes of the treatment group will be compared with the changes of the placebo group to illustrate the treatment effect of Lycium Barbarum
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Lycium Barbarum | Placebo
Number analyzed (Participants) | 23 | 19
dB | 0.32 (2.93) | -0.16 (0.94)

3. Secondary Outcome: Amplitudes of Flash Electroretinogram
Description: The cone responses from electroretinogram will be measured at the time point of baseline and 12 months. The cone response is related to the activity of the cone photoreceptor under light stimulation.
  The change of cone response b-wave amplitude (uV) between 12-month and baseline will be provided to show the effect of interventions. The b-wave amplitude is to measure the magnitude of electrical responses of cone cells in the retina.
  The changes of the treatment group will be compared with the changes of the placebo group to illustrate the treatment effect of Lycium Barbarum.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: uV
Arm/Group | Lycium Barbarum | Placebo
Number analyzed (Participants) | 23 | 19
uV | 2.75 (9.17) | -4.00 (7.38)

4. Secondary Outcome: Implicit Times of Flash Electroretinogram
Description: The cone responses from electroretinogram will be measured at the time point of baseline and 12 months. The cone response is related to the activity of the cone photoreceptor under light stimulation.
  The change of cone response b-wave implicit time (ms) between 12-month and baseline will be provided to show the effect of interventions. The b-wave implicit time is to measure the physiological changes of cone cells in the retina.
  The changes of the treatment group will be compared with the changes of the placebo group to illustrate the treatment effect of Lycium Barbarum.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Lycium Barbarum | Placebo
Number analyzed (Participants) | 23 | 19
msec | -1.33 (5.03) | -1 (6.69)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Self reporting
Arm/Group | Lycium Barbarum | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/19
Other Adverse Events (participants affected / at risk) | 0/23 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No